CLINICAL TRIAL: NCT00836225
Title: A Phase I , Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ISIS 388626 Administered to Healthy Volunteers
Brief Title: Safety, Tolerability and Activity Study of Multiple Doses of ISIS-SGLT2Rx in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 388626-CS1
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; SGLT2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ISIS 388626

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- A (Experimental): 50 mg ISIS 388626 vs Placebo, s.c. injection
  Interventions: Drug: ISIS 388626
- B (Experimental): 100 mg ISIS 388626 vs Placebo, s.c. injection
  Interventions: Drug: ISIS 388626
- C (Experimental): 200 mg ISIS 388626 vs Placebo, s.c. injection
  Interventions: Drug: ISIS 388626
- D (Experimental): 400 mg ISIS 388626 vs Placebo, s.c. injection
  Interventions: Drug: ISIS 388626
- AA (Experimental): 50 mg ISIS 388626, 3x over 1 week s.c. injection, weekly s.c. injection for 5 weeks vs Placebo
  Interventions: Drug: ISIS 388626
- BB (Experimental): 100 mg ISIS 388626, 3x over 1 week s.c. injection, weekly s.c. injection for 5 weeks vs Placebo
  Interventions: Drug: ISIS 388626
- AAA (Experimental): 50 mg ISIS 388626, weekly s.c. injection for 13 weeks vs Placebo
  Interventions: Drug: ISIS 388626
- BBB (Experimental): 100 mg ISIS 388626, weekly s.c. injection for 13 weeks vs Placebo
  Interventions: Drug: ISIS 388626
- CCC (Experimental): 200 mg ISIS 388626, weekly s.c. injection for 13 weeks vs Placebo
  Interventions: Drug: ISIS 388626
- FFF (Experimental): 50 mg ISIS 388626, weekly s.c. injection for 13 weeks vs Placebo
  Interventions: Drug: ISIS 388626

INTERVENTIONS:
Drug: ISIS 388626 — 4 arms of single dose s.c. injections: A 50 mg, B 100 mg, C 200 mg, D 400 mg, 2 arms of multi-dose: 3 s.c. injections over 1 week followed by 5 weekly s.c. injections: AA 50 mg, BB 100 mg 3 arms of multi-dose 13 weekly s.c. injections: AAA 50 mg, BBB 100 mg, CCC 200 mg, FFF 50 mg
  Placebo: 0.9% sterile saline

SUMMARY:
The primary purpose of this trial is to assess the safety and tolerability of ISIS-SGLT2Rx when given at increasing single doses and to assess the safety and tolerability of the same doses when given multiple times.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of a single subcutaneous injection of ISIS-SGLT2Rx administered at four increasing dose levels (50, 100, 200, 400 mg) and to evaluate the safety and tolerability of multiple doses of ISIS 388626 administered subcutaneously of either 6 or 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Male or female gender although females must be post-menopausal or surgically sterile (hysterectomy, oophorectomy or tubal ligation)
* Give written informed consent to participate in the study and availability for all study requirements
* Fasting plasma glucose </= the upper limit of the laboratory's reference range (ULN)
* HbA1c </= ULN
* BMI < 30 kg/m²
* Agree to maintain steady hydration throughout study participation and agree not to fluid restrict

Exclusion Criteria:

* Pregnant women, nursing mothers or women of childbearing potential
* Clinically significant abnormalities in medical history or physical examination
* Clinically significant abnormalities in laboratory examination (including ALT > ULN, AST > ULN, bilirubin > ULN, creatinine > ULN, urine protein positive by urine dipstick, platelets < lower limit of normal and any other clinically significant laboratory findings)
* Estimated GFR < 60 mL/min per 1.73m²
* History of clinically significant abnormalities in coagulation parameters
* Positive test result for HIV, hepatitis B virus, and/or hepatitis C virus
* Active infection requiring antiviral or antimicrobial therapy
* Subjects on chronic or acute prescription medication may be permitted after discussion with the Isis Medical Monitor
* Malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for > 1 year)
* Any other concurrent condition which, in the opinion of the Investigator, would preclude participation in this study or interfere with compliance
* Past and present history of alcohol or drug abuse (defined as > 3 units daily)
* Undergoing or have undergone treatment with another investigational drug, biologic agent or device within 90 days prior to Screening
* Blood donation within three months of Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple doses of ISIS-SGLT2Rx administered subcutaneously | 30 days for single dose, 11 weeks for 6-week dosing, 18 weeks for 13-week dosing

SECONDARY OUTCOMES:
Pharmacokinetic profile all doses and Pharmacodynamics for multi-dose groups | 3 days for single dose, 11 weeks for 6-week dosing, 18 weeks for 13-week dosing

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cohen, MD, PhD, Principal Investigator — Center for Human Drug Research
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Tekendo-Ngongang C, Gleeson JG, Mignon L. Treating the Untreatable: Antisense Oligonucleotides as an Individualized Therapy for Rare Genetic Kidney Diseases. J Am Soc Nephrol. 2024 Dec 1;35(12):1774-1777. doi: 10.1681/ASN.0000000532. Epub 2024 Sep 27. No abstract available. PMID 39331470